CLINICAL TRIAL: NCT05093920
Title: Role of Drug Eluting Bead Transarterial Chemoebolization Versus Conventional Transarterial Chemoembolization in Treatment of Hepatocellular Carcinoma
Brief Title: Role of DEB-TACE Versus c-TACE in Treatment of HCC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Elsaman Mohamed, Assistant Lecturer at department of diagnostic and interventional radiology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-10-31
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug Eluting Bead Transarterial Chemoembolization (Active Comparator): Drug Eluting Bead Transarterial Chemoembolization
  Interventions: Drug: Doxorubicin-Eluting Beads
- conventional Transarterial Chemoembolization (Active Comparator): conventional Transarterial Chemoembolization
  Interventions: Drug: Doxorubicin-Eluting Beads

INTERVENTIONS:
Drug: Doxorubicin-Eluting Beads — * The patients will be categorized in two randomized groups; c-TACE group (A) and DEB-TACE group (B).
  * After patient counseling and obtaining a written consent to participate in the study, both groups will be subjected to the interventional procedure according to patient group; Group A; Lipidol-Doxorubicin emulsion material followed by gel foam embolic material will be injected through the catheter directly into tumor feeding vessels through transarterial catheter.
  Group B; Doxorubicin-Eluting Beads will be injected through the catheter directly into tumor feeding vessels through transarterial catheter.
  Other Names: Lipidol-Doxorubicin emulsion

SUMMARY:
Hepatocellular carcinoma (HCC) is listed as the sixth most common cancer worldwide and the third most frequent cause of cancer-related mortality. The majority of HCC cases occurs stem from chronic liver disease and cirrhosis.

Hepatocellular carcinoma accounts for approximately 70% to 90% of all primary liver cancers. Trans-arterial Chemoembolization is the most widely utilized and is considered the first-line treatment recommended for patients staged as intermediate HCC (Barcelona Clinic Liver Cancer stage B). If applied correctly, TACE can produce survival benefits without adversely affecting hepatic functional reserve.

Two TACE techniques have been used since 2004, conventional TACE (c-TACE) and TACE with drug-eluting beads (DEB-TACE). Conventional TACE was evidenced first to treat intermediate stage HCC patients.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is listed as the sixth most common cancer worldwide and the third most frequent cause of cancer-related mortality. The majority of HCC cases occurs stem from chronic liver disease and cirrhosis.

Hepatocellular carcinoma accounts for approximately 70% to 90% of all primary liver cancers. HCC patients have been suffering from poor prognosis with 5-year survival being roughly 10% to 15% for decades despite the progress in screening, diagnosis, and treatment, which is mainly resulted from that most patients are already in the moderate or advanced stage at diagnosis, whom can only receive palliative treatments.

At the level of the individual patient, concomitant cirrhosis and the number, size, and location of hepatocellular tumors will affect the treatment approach. In addition, multiple disease-related factors need to be taken into account, such as the presence of vascular involvement or extra-hepatic disease, when deciding on the best treatment options for these patients. Consequently, a multidisciplinary approach involving several physicians with different specialties (e.g., diagnostic and interventional radiologists, surgical oncologists, hepatologists, and medical oncologists) is necessary to determine the best approach to treatment and maximize potential outcomes for patients with HCC.

The liver has a dual vascular supply via the hepatic artery and the portal vein. The rationale of the trans-arterial embolotherapies is explained by the fact that liver malignancies are predominantly supplied by the hepatic artery, which allows delivering the chemotherapy directly to the tumor-feeding artery while sparing the healthy hepatic tissue mainly supplied by the portal vein.

Loco regional treatments are a set of therapeutic approaches that directly target tumors in the liver. Among the loco regional modalities, trans-arterial chemoembolization (TACE) involves the local delivery of chemotherapy to the tumor and is generally recommended for patients with liver-limited disease. Several randomized trials have been conducted to examine the efficacy and safety of TACE.

According to the Barcelona Clinic Liver Cancer (BCLC) staging system, TACE is the first-line treatment for patients with intermediate stage HCC, including those with large or multinodular HCC, well-preserved liver function, and no cancer-related symptoms or evidence of vascular invasion or extrahepatic spread. Recent advances allow TACE treatment of both early stage patients (i.e. those with a solitary nodule or up to 3 nodules under 3 cm) and some advanced stage patients.

Trans-arterial Chemoembolization is the most widely utilized and is considered the first-line treatment recommended for patients staged as intermediate HCC (Barcelona Clinic Liver Cancer stage B). If applied correctly, TACE can produce survival benefits without adversely affecting hepatic functional reserve.

Two TACE techniques have been used since 2004, conventional TACE (c-TACE) and TACE with drug-eluting beads (DEB-TACE). Conventional TACE was evidenced first to treat intermediate stage HCC patients. It combines the trans-catheter delivery of chemotherapy using Lipiodol-based emulsion plus an embolizing agent to achieve strong cytotoxic and ischemic effects. Drug-eluting beads (DEB) were developed in order to slowly release chemotherapeutic agents, and to increase ischemia intensity and duration.

The introduction of TACE with drug eluting beads (DEB-TACE) was primarily developed to enhance the delivery of the chemotherapeutic agent while minimizing systemic toxicity and to provide a standardized embolizing effect. DEBs are embolic microspheres loaded with a chemotherapeutic agent (mostly doxorubicin) with the ability of slow drug release, which should ensure high local and low systemic drug concentrations. Indeed, systemic levels of doxorubicin were significantly lower in patients receiving DEB-TACE compared to patients receiving c-TACE with Lipiodol.

DEB-TACE was introduced 10 years ago with the aim to improve the overall c-TACE outcomes and to diminish the side effects of the procedure. It is based on the use of microspheres that exploit ionic bonds and are able to actively sequester and then slowly release the cytotoxic drug inside the target lesion. Moreover, the use of particles allows a deeper distal embolization of small vessels, ensuring a permanent highly selective occlusion of the tumor-feeding arteries.

DEB-TACE has several advantages over c-TACE, such as the delivery of higher concentrations of chemotherapeutic agents directly to tumors, lower rates of systemic complications, greater efficacy in advanced stage or large tumors, and better standardization of the procedure itself.

ELIGIBILITY:
Inclusion Criteria:

* - Child-Pugh A or B cirrhosis.
* ECOG performance status (PS) Grade 2 or below.
* BCLC stage B or C.
* No serious concurrent medical illness.
* Radiologically or histologically proven HCC (an alpha-fetoprotein level > 500 ug/ml in the presence of radiological findings suggestive of HCC in a patient with chronic HBV or HCV infection is considered eligible).
* Unresectable and locally advanced disease without extra-hepatic disease.
* Nodular tumor morphology with measurable lesion on CT with less than 50% involvement of liver by HCC.
* Size of largest tumor is less than or equal to 15cm in largest dimension.
* Number of main tumor is less than or equal to 5, excluding associated small satellite lesions.
* Patent main portal vein.

Exclusion Criteria:

* - Child-Pugh C cirrhosis (evidence of poor liver function).
* History of significant concurrent medical illness such as ischemic heart disease or heart failure.
* Serum creatinine level > 2 mg/dL.
* Presence of extrahepatic metastasis.
* Predominantly infiltrative lesion.
* Diffuse tumor morphology with extensive lesions involving both lobes.
* Hepatic artery thrombosis.
* Thrombosis of the main portal vein.
* Tumor invasion of portal branch of contralateral lobe.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Tumor size | four-six weeks after treatment
  Triphasic CT scan of the liver measures the maximum diameter of tumor according to modified RECIST (mRecist) criteria.

SECONDARY OUTCOMES:
Serum Alpha-fetoprotein level ng/ml. | four-six weeks after treatment
  Laboratory test of Serum alpha-fetoprotein level (AFP) ng/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed E Mohamed, Master, Principal Investigator — Sohag University; Mohamed Z Ali, MD, Study Chair — Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho SM, Chu HH, Kim JW, Kim JH, Gwon DI. Initial Transarterial Chemoembolization (TACE) Using HepaSpheres 20-40 microm and Subsequent Lipiodol TACE in Patients with Hepatocellular Carcinoma > 5 cm. Life (Basel). 2021 Apr 18;11(4):358. doi: 10.3390/life11040358. PMID 33919658
- [Background] Gholam PM, Iyer R, Johnson MS. Multidisciplinary Management of Patients with Unresectable Hepatocellular Carcinoma: A Critical Appraisal of Current Evidence. Cancers (Basel). 2019 Jun 22;11(6):873. doi: 10.3390/cancers11060873. PMID 31234476
- [Background] Li H, Wu F, Duan M, Zhang G. Drug-eluting bead transarterial chemoembolization (TACE) vs conventional TACE in treating hepatocellular carcinoma patients with multiple conventional TACE treatments history: A comparison of efficacy and safety. Medicine (Baltimore). 2019 May;98(21):e15314. doi: 10.1097/MD.0000000000015314. PMID 31124925
- [Background] Melchiorre F, Patella F, Pescatori L, Pesapane F, Fumarola E, Biondetti P, Brambillasca P, Monaco C, Ierardi AM, Franceschelli G, Carrafiello G. DEB-TACE: a standard review. Future Oncol. 2018 Dec;14(28):2969-2984. doi: 10.2217/fon-2018-0136. Epub 2018 Jul 10. PMID 29987957